CLINICAL TRIAL: NCT02316262
Title: Targeted Reinnervation for Neuromas as a Means to Improve Prosthesis Control in Major Limb Amputation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Gregory Dumanian, Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TR Prosthetic Control
Record Dates: First submitted 2014-12-10; First posted 2014-12-12 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Neuroma; Pain; Prosthesis User; Prosthesis Failure
MeSH Terms: conditions — Neuroma; Pain; Prosthesis Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TR (Experimental): All subjects enrolled in this study will undergo pre-operative evaluation, anesthesia, and dissection to identify the painful residual limb neuroma(s). Gentle traction will be applied to the nerve while excising the neuroma (traction neurectomy) allowing the nerve to retract more proximally.Targeted muscle reinnervation involves transfer of residual nerves to otherwise redundant target muscles. Native motor innervation of the target muscle is cut, and the residual nerves-after excision of end-neuromas-are coapted to the motor end point of the motor nerve, close to its point of entry into the muscle.
  Interventions: Procedure: Targeted Muscle Reinnervation

INTERVENTIONS:
Procedure: Targeted Muscle Reinnervation — Targeted reinnervation (TR) is a surgical procedure originally designed to provide intuitive control of upper limb prostheses through transfers of residual nerves to otherwise redundant target muscle. Native motor innervation of the target muscle is cut, and the residual nerves-after excision of end-neuromas-are coapted to the motor end point of the motor nerve, close to its point of entry into the muscle. The central principle underlying the nerve transfers in TR surgery is to reestablish the function of the amputated nerve and allow intuitive, seamless prosthesis control.
  Other Names: Targeted Reinnervation

SUMMARY:
Subjects are being asked to participate in this study because they have an arm or leg amputation and have developed pain related to a neuroma (an ongoing localized pain related to a cut nerve ending).

The investigators are studying how targeted reinnervation (TR) helps to both treat neuroma pain and to have increased prosthetic control. This surgery connects these cut nerve endings to nerves going into nearby nonfunctional muscles. This surgery was developed to allow amputees to have better prosthesis control. By chance, neuroma pain improved significantly with TR. The investigators, therefore, are conducting this clinical trial. The investigators will ask all participants to fill out a questionnaire both before and after surgery. This will help us understand how a neuroma affects the quality of life of amputee will allow us to understand how to best improve neuroma pain and prosthesis control.

In order to confirm the presence and location of the neuroma before surgery, a magnetic resonance image (MRI) will be performed. Taking these pictures requires subjects to lie still for a short period of time but does not involve any invasive procedures.

DETAILED DESCRIPTION:
Loss of an arm or leg is a significant injury that affects a person's job prospects, personal relationships, and overall quality of life. Approximately 25% of all amputees will develop chronic local pain in the remaining part of their amputated limb. This pain is caused by neuromas- disorganized nerve endings and scar tissue that form when an injured nerve tries to heal. Every cut nerve will develop a neuroma unless the two ends of the nerve can be rejoined. With limb amputation, the nerves are cut and one end is lost with the limb, preventing the nerve from repairing itself. Instead, the cut nerve ending forms a painful neuroma. Chronic pain from neuromas is a major reason that amputees cannot wear or use their prostheses comfortably and increases their disability.

Even when a limb is amputated, the nerves that used to control that limb still carry messages from the brain. Those messages are intended to tell the muscles how or when to move the missing limb, but after amputation, these limb-control nerves are no longer connected to muscles. In 2002, researchers at Northwestern Memorial Hospital in conjunction with the Rehabilitation Institute of Chicago developed a new type of surgery called targeted muscle reinnervation (TMR). In TMR, limb-control nerves are transferred so that they can control new target muscles. The neuromas from the limb-control nerves are removed, then the small nerve that controls the target muscle is cut. The two nerves are joined together so that the limb-control nerve can then grow into, or reinnervate the target muscle. After TMR, when the person tries to move the missing limb, the target muscle contracts instead and these signals can be detected and used to control a prosthesis. TMR has now been done successfully almost 100 times worldwide. Interestingly, almost all of the patients who had painful neuromas before TMR had no neuroma pain after surgery. This result was investigated in laboratory studies - both rat and rabbit amputee neuromas were "cured" with TMR. We think that giving the cut nerve endings somewhere to go and something to do prevents a neuroma from forming.

We will measure the effectiveness of both surgeries using an internet-based amputee pain questionnaire. We expect that TMR will be more effective for neuroma pain and prosthesis control than the standard treatment. This will change how patients with neuroma pain are treated and help thousands of patients with amputations.

ELIGIBILITY:
Inclusion Criteria:

* Adult, 18 years or older: the Patient Reported Outcomes Measurement Information System (PROMIS) questionnaire is not validated for pain-related evaluation in minors
* An upper limb amputation above the wrist with or without a residual limb or a lower limb amputation above the ankle with a residual limb
* A neuroma within the residual limb: defined as patient-reported chronic localized pain consistent with a physical exam that demonstrates that the pain is related to a cut nerve and excludes other causes. There must be a supporting Tinel's sign on physical exam, or localization of a neuroma by prior intervention (surgical or otherwise) to distinguish the pain from phantom limb pain or cold intolerance that are nonspecific signs of nerve damage that would not be affected by treatment of a neuroma
* English or Spanish speaking

Exclusion Criteria:

* Prior TR Surgery: these patients have already had a procedure to improve their prosthetic function and in these cases the nerves have been shortened. To perform a second TR procedure with the previously shortened nerves would require a significant proximal dissection and potentially greater soft tissue morbidity than the standard treatment.
* Cognitive impairment, due to TBI or other causes, sufficient to adversely affect understanding of or compliance with study requirements, ability to respond to questionnaires, or ability to give informed consent: The ability to understand and comply with requirements of the study is essential in order for the study to generate useable, reliable data. The ability to obtain relevant feedback through questionnaires is essential to this study.
* Pre-operative assessment that precludes the patient from being eligible for TR or control surgery due to technical surgical concerns.
* Significant other comorbidity: Any other medical issues or injuries that would preclude safe administration of anesthesia or surgical intervention.
* Participation in other ongoing studies related to neuropathic pain.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-10; Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Improvement in pain of the amputated limb after surgery (survey results) | 12 months
  Compare patient-reported pre-operative survey results to those after surgical intervention at intervals over time (1 month, 3 months,6 months, 9 months,1 year, and then every six months thereafter until the conclusion of the study).
Improvement in physical functioning (prosthesis wear and function), after surgery | 12 months
  Using the same PROMIS platform, general health, physical functioning (including functional prosthesis wear), and satisfaction following surgery will also be assessed as important secondary outcomes, resulting in a more comprehensive and objective understanding of the effects of the two surgical approaches on neuroma pain.
  Another particularly useful tool for this study is the Orthotics and Prosthetics User Survey (OPUS) Functional Status. The OPUS is a validated instrument that assesses how well patients are using their prostheses. Thus, we will examine a very important secondary measure of neuroma pain-the ability to use a prosthesis. Prosthesis use is often the primary problem for individuals with painful neuromas; they hurt most during walking with a prosthesis or when wearing a prosthetic arm.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Northwestern University, Chicago, Illinois
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - The Ohio State University, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - San Antonio Military Medical Center, San Antonio, Texas